CLINICAL TRIAL: NCT01874483
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 187004 CL in Patients With Type 2 Diabetes Mellitus (Randomized, Double-blind Placebo-controlled Within Dose Groups)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Doses of BI 187004 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1307.2; 2013-000312-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (8):
- BI 187004 dose 1 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 187004
- BI 187004 dose 2 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 187004
- BI 187004 dose 3 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 187004
- BI 187004 dose 4 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 187004
- BI 187004 dose 5 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 187004
- BI 187004 dose 6 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 187004
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- BI 187004 dose 7 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 187004

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: Placebo
Drug: BI 187004 — BI 187004, dose 2
  Arms: BI 187004 dose 2
Drug: BI 187004 — BI 187004, dose 4
  Arms: BI 187004 dose 4
Drug: BI 187004 — BI 187004, dose 5
  Arms: BI 187004 dose 5
Drug: BI 187004 — BI 187004, dose 6
  Arms: BI 187004 dose 6
Drug: BI 187004 — BI 187004, dose 7
  Arms: BI 187004 dose 7
Drug: BI 187004 — BI 187004, dose 1
  Arms: BI 187004 dose 1
Drug: BI 187004 — BI 187004, dose 3
  Arms: BI 187004 dose 3

SUMMARY:
To investigate safety, tolerability, pharmacokinetics and pharmacodynamics of BI 187004 following multiple dose administration over 14 days.

ELIGIBILITY:
Inclusion criteria:

1. Type 2 diabetes mellitus
2. Current treatment with no more than one anti-diabetic drug (except for insulin and GLP-1 analogues)
3. Males or post-menopausal or surgically sterilised females
4. Age from 20 and to 70 years
5. HbA1c less or equal to 8.5%
6. BMI 28-40 kg/m2
7. Subjects must be able to understand an comply with study requirements

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal that the investigator considers to be of not acceptable clinical relevance
2. Repeated measurement of systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 95 mm Hg
3. Myocardial infarction, stroke or transient ischemic attack within 6 months prior to informed consent
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders besides type 2 diabetes, hyperlipidaemia or medically treated hypertension
5. Surgery of the gastrointestinal tract that might affect absorption and elimination of the study drug
6. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or relevant neurological disorders besides polyneuropathy
7. Chronic or relevant acute infections (e.g. HIV, hepatitis)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | up to 15 days postdose

SECONDARY OUTCOMES:
AUCt,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval t after administration of the first dose) | up to 8 days postdose
Cmax t,1 (maximum measured concentration of the analyte in plasma after administration of the first dose) | up to 8 days postdose
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) | up to 8 days postdose
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) | up to 8 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1307.2.1 Boehringer Ingelheim Investigational Site, Neuss, Germany

REFERENCES:
- [Derived] Bianzano S, Schepers C, Wolff M, Heise T, Plum-Moerschel L. Selective Inhibition of 11beta-Hydroxysteroiddehydrogenase-1 with BI 187004 in Patients with Type 2 Diabetes and Overweight or Obesity: Safety, Pharmacokinetics, and Pharmacodynamics After Multiple Dosing Over 14 Days. Exp Clin Endocrinol Diabetes. 2022 Dec;130(12):773-782. doi: 10.1055/a-1932-3136. Epub 2022 Nov 7. PMID 36343645